CLINICAL TRIAL: NCT00223457
Title: Factors That Influence Compliance With Disease-Modifying Therapy in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Biogen (Industry)
Other Study IDs: MS DMA Compliance
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2007-01-25 (Estimated); Status verified 2005-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; compliance; adherence; disease modifying therapy; depression; hope; quality of life
MeSH Terms: conditions — Multiple Sclerosis; Patient Compliance; Depression

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: Factors that influence compliance

SUMMARY:
The purpose of this study is to evaluate the coorelation between patient factors, health care provider factors, drug factors and compliance in patients with relapsing forms of multiple sclerosis (RMS) treated with Disease Modifying Agents (DMA). We hypothesize that a number of factors influence compliance with DMA's.

DETAILED DESCRIPTION:
While compliance rates with interferons and glatiramer acetate treatment have been high when assessed in the context of controlled clinical trials, we have observed substantially less consistent rates of drug administration in general practice. Correspondingly, the magnitude of drug efficacy achieved on clinical and surrogate markers of disease activity in the latter patient group may be compromised compared to patients participating in controlled clinical trials. Further, in many circumstances, the perception of breakthrough disease simply constitutes treatment noncompliance.

The National Multiple Sclerosis Society reports only 50% of all MS patients and 60% with relapsing remitting MS are taking disease modifying agents in the U.S. (Zwibel 2003) A number of studies have investigated this challenging issue. When glatiramer acetate therapy was specifically evaluated, the investigators found several factors to be associated with compliance. They discovered adherence to be higher with the patient perception of physician support of the medication prescribed, patient sense of control, higher levels of hope and no previous use of other disease modifying therapy (Fraser, Hadjimichael, and Vollmer 2001). Another study by Hadjimichael and Vollmer (1999) surveyed patients for reasons that medications were discontinued. Disease progression, lack of improvement and side effects were some of the reasons reported by patients for stopping disease-modifying therapy.

Depression is another factor found to impact adherence. Mohr, Goodkin, Likosky, Gatto, Baumann and Rudick (1997) saw increased rates of compliance with Interferon beta-1b therapy in multiple sclerosis with the treatment of underlying depression. The study showed that patients with increased depression were more likely to discontinue therapy. This link of depression has also been demonstrated with noncompliance with antihypertensive medications. (Wang,Bohn, Harooni et al. 2002) In another study, Mohr (2001) saw patient's experienced level of anxiety with their injections was related to adherence.

We hypothesize that a number of factors influence compliance with DMA's, these include:

1. Patient factors

   1. Perceived quality of life
   2. Empowerment, sense of control & hope
   3. Support structure (family, faith, injection assistance, etc.)
   4. Depression
   5. Fatigue
   6. Cognitive problems
   7. Perception of drug efficacy (benefit over costs)
2. Physician (HCP support) factors

   1. Patient's perception of MD support
   2. Relationship with MD
   3. Access to nurses and other HCP support functions
   4. Services provided by physician/clinical practice (i.e. academic, community-based, or MS clinic)
   5. Adequate education on MS, establishing reasonable expectations concerning the benefit derived from therapy,
3. Drug factors

   1. complexity of drug administration
   2. drug associated side effects/tolerability
   3. Perceived MS symptom control
   4. Insurance coverage of the injection
   5. Concomitant medications

Once the factors that contribute to noncompliance to DMA therapies are identified, healthcare professionals can evaluate how they can be impacted. The healthcare team can work towards addressing those barriers where there is a possibility for change, to help improve patient outcomes.

The primary objective of this study is to evaluate the correlation between patient factors, HCP support factors, drug factors, and compliance in patients with relapsing forms of multiple sclerosis (RMS) treated with Disease Modifying Agents (DMA).

The secondary objectives of the study are to determine differences in patient compliance between patients treated by academic centers/MS specialists and community neurology centers; and to determine the factors that impact this difference.

Patients are asked to sign (electronic agreement) a consent to participate in this confidential study when they initially log-on to the study website. Patients are assigned a unique identification number when they log into the internet for the first time to complete the study survey. By using this assigned number, health information will be protected for each individual. Patient names will be used only for purposes of check distribution and participation in following studies if the patient consents. If a patient drops out of the study, TNS Healthcare will contact the patient to find out the reason. The treating physician does not know who elected to participate in the study.

Study Design- This is a multicenter, retrospective trial administered through patient surveys. We are utilizing the validated MS quality of life 54 (MSQOL-54), the Beck's Fast Screen for medical patients, the Hope Herth Index, and a patient self-reported drug compliance survey. The participating neurologists were asked to give patients with relapsing forms of MS flyers describing the study. The flyers direct patients to the designated study website to complete the confidential survey by internet. As described below, patients log-on to the website a total of 3 times during the study period, Baseline (time 0), Month 1 (Time 1) and Month 2 (Time 2). Patients log on with a unique identification number rather than names to ensure that confidentiality is maintained throughout the study.

The goal is to have an equal number of patients treated with the four different DMA's, AVONEX, Rebif, Copaxone, and Betaseron. The sample is to include at least 150-200 patients from each of the MS Centers and 15-20 patients from each of the community sites, for a total of approximately 1040 patients. Power analysis was performed assuming a 15% critical effect value. The sample size was calculated to provide 80% power to detect the critical effect value at a confidence interval of 95%. Response rates are estimated to be 60% for the first wave and 75% for the second wave of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing form of multiple sclerosis
* Age 18 or older
* Therapy with disease modifying agent (Glatiramer acetate, Interferon Beta-1b, ot Interferon Beta 1a (IM or SC) for at least 6 months
* Access to the internet to complete the study survey

Exclusion Criteria:

* Diagnosis of progressive forms of multiple sclerosis
* Therapy on DMA for less than 6 months
* Inability to complete the survey
* Participation in other investigational studies within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040
Dates: Start 2004-04; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Elliot M Frohman, MD, PhD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Katherine D Treadaway, LCSW, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] 1. Zwibel, H. Practical Issues in MS Clinical Management, Patient Choice, Safety, and Adherence. International Journal of MS Care 2003 Oct: (suppl) 18-21.
- [Background] Fraser C, Hadjimichael O, Vollmer T. Predictors of adherence to Copaxone therapy in individuals with relapsing-remitting multiple sclerosis. J Neurosci Nurs. 2001 Oct;33(5):231-9. doi: 10.1097/01376517-200110000-00003. PMID 11668881
- [Background] Hadjimichael O, Vollmer T. Adherence to injection therapy in multiple sclerosis:patients survey. Neurology 1999; 52 (suppl 2):A549
- [Background] Mohr DC, Boudewyn AC, Likosky W, Levine E, Goodkin DE. Injectable medication for the treatment of multiple sclerosis: the influence of self-efficacy expectations and injection anxiety on adherence and ability to self-inject. Ann Behav Med. 2001 Spring;23(2):125-32. doi: 10.1207/S15324796ABM2302_7. PMID 11394554
- [Background] Mohr DC, Goodkin DE, Likosky W, Gatto N, Baumann KA, Rudick RA. Treatment of depression improves adherence to interferon beta-1b therapy for multiple sclerosis. Arch Neurol. 1997 May;54(5):531-3. doi: 10.1001/archneur.1997.00550170015009. PMID 9152109
- [Background] Wang PS, Bohn RL, Knight E, Glynn RJ, Mogun H, Avorn J. Noncompliance with antihypertensive medications: the impact of depressive symptoms and psychosocial factors. J Gen Intern Med. 2002 Jul;17(7):504-11. doi: 10.1046/j.1525-1497.2002.00406.x. PMID 12133140
- [Result] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530